CLINICAL TRIAL: NCT00750815
Title: An Open Label Phase I/II Study of the Safety and Efficacy of Cyclophosphamide, Bortezomib (VELCADE), Pegylated Liposomal Doxorubicin (DOXIL), and Dexamethasone, (CVDD) in Newly Diagnosed Patients With Multiple Myeloma
Brief Title: Cyclophosphamide, VELCADE, DOXIL, and Dexamethasone, (CVDD) in Newly Diagnosed Patients With Multiple Myeloma (MM)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Ortho Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15399; 106692 (Other: USF IRB); Millennium X05248 (Other: Millennium Pharmaceuticals, Inc.); DOXILMMY2008 (Other: Ortho Biotech, Inc.)
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Results first posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2013-09

CONDITIONS: Multiple Myeloma
Keywords: B Cell; hematologic malignancy; plasma; bone marrow
MeSH Terms: conditions — Multiple Myeloma; Hematologic Neoplasms | interventions — Cyclophosphamide; Bortezomib; liposomal doxorubicin; Dexamethasone; 1-dodecylpyridoxal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A. Phase I - Dose Escalation (Experimental): Dose of Cyclophosphamide to depend on how many patients we treated:
  * Dose Level 1: Cyclophosphamide 250 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Dose Level 2: Cyclophosphamide 500 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Dose Level 3: Cyclophosphamide 750 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Dose Level 4: Cyclophosphamide 750 mg /m^2 IV Day 1; VELCADE, 1.3 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  Interventions: Drug: Cyclophosphamide; Drug: Bortezomib; Pegylated Liposomal Doxorubicin; Dexamethasone (VDD)
- B. Phase II - Maximum Planned Dose (MPD) (Experimental): Participants received Cyclophosphamide and VELCADE at Level 4 (the MPD) at the same schedule of the Phase I study. Pegylated doxorubicin and Dexamethasone were given at the same doses and schedule as the Phase I part of study.
  Interventions: Drug: Cyclophosphamide; Drug: Bortezomib; Pegylated Liposomal Doxorubicin; Dexamethasone (VDD)

INTERVENTIONS:
Drug: Cyclophosphamide — Enroll patients into 4 different dose levels. The dose of Cyclophosphamide they receive will depend on how many patients have been treated.
  Other Names: Cytoxan
Drug: Bortezomib; Pegylated Liposomal Doxorubicin; Dexamethasone (VDD) — Patients will receive Bortezomib, Pegylated Liposomal Doxorubicin and Dexamethasone at standard doses.
  Other Names: VELCADE; DOXIL®; PLD; CVDD; VDD

SUMMARY:
Cyclophosphamide is a chemotherapy agent with known activity in myeloma. The new regimen that we will test in this study is called CVDD and contains Cyclophosphamide with Bortezomib (VELCADE), Pegylated Liposomal Doxorubicin (DOXIL®, PLD), and Dexamethasone (VDD).

The purpose of this study is to determine if the addition of another type of chemotherapy agent, Cyclophosphamide, to the regimen VDD (CVDD) is well tolerated and improves response rates in myeloma. We will also find the highest safe dose of the study drugs taken together that a patient can tolerate, and how long it takes for multiple myeloma patients to respond after they have taken the study drugs and how long the response lasts.

DETAILED DESCRIPTION:
The first cohort of 3 participants enrolled into Phase I of the study will receive dose level 1. A full safety evaluation will be conducted when these participants have completed one cycle (21 days) of combination therapy. Further patient accrual will be suspended while the safety data is evaluated at each dose level.

Dose escalation for subsequent patients will proceed through dose levels 2, 3 and 4 as follows:

* If no dose limiting toxicity (DLT) is reported in the first 3 participants at a dose level, that dose level will be considered safe and 3 participants will be enrolled at the next dose level. If 1/3 participants in a cohort at a dose level has a DLT, the dose level will be expanded to obtain 6 evaluable participants.
* If > 1 of 3 participants in a cohort experience DLT, that dose level will not be considered safe. No further dose escalation will take place, and the immediate lower dose level will be considered the maximum planned dose (MPD) if 6 patients had been enrolled at that dose level. Otherwise, expand the immediate lower dose level to 6 evaluable patients*.
* If there are < 2 participants with a DLT among the expanded cohort of 6 evaluable participants, a cohort of 3 participants will be enrolled in the next higher dose level.
* If there are 2 or more participants with a DLT among the expanded cohort of 6 evaluable participants, that dose level will not be considered safe. No further dose escalation will take place, and the immediate lower dose level will be considered the MPD if 6 patients had been enrolled at that dose level. Otherwise, expand the immediate lower dose level to 6 evaluable patients*.
* * If DLT occurs in no more than 1 patient in the expanded dose cohort, then that dose level will be considered MPD. Otherwise, the dose will be further de-escalated in a similar fashion until the MPD is reached.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign informed consent form; equal to or greater than 18 years of age at time of consent
* Able to adhere to the study visit schedule and other protocol requirements
* Diagnosed active multiple myeloma
* Measurable myeloma paraprotein levels in serum (≥ 0.5 g/dL) or urine (≥ 0.2 g excreted in a 24-hour urine collection sample), or serum involved free light chains ( >10mg/dl) provided that the k/l ratio is abnormal
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Performance status of 3 allowed if related to bony disease.
* Bilirubin ≤ 1.5x upper limits of normal (ULN)
* Liver enzymes: alanine transaminase (ALT)or aspartic transaminase (AST) ≤ 2.5 x ULN. In the presence of liver metastases, AST / ALT, alkaline phosphatase and total bilirubin must not exceed 3x upper limit of normal (i.e.: must be ≤ 3x ULN).
* Adequate bone marrow function:
* Absolute neutrophil count (ANC) ≥ 1,000 cells/mm³ (1.0 x 10^9/L). Patients with bone marrow >50% plasma cells are permitted to have a neutrophil count of < 1,000 cells/mm³.
* Platelets ≥ 100,000 cells/mm³. Patients with bone marrow >50% plasma cells are permitted to have a Platelet count ≤ 100, 000 cells/mm³
* Hemoglobin > 8 g/dL (transfusion allowed to increase the Hgb)
* Adequate renal function: Creatinine ≤ 2.5 mg/dL
* Must have 2-d echocardiogram or multigated acquisition (MUGA) scan indicating left ventricular ejection fraction (LVEF) ≥ 50% within 42 days prior to first dose of study drug. A MUGA scan or 2- d Echocardiogram may be used, but the same test must be used throughout study) to evaluate LVEF.
* Women of childbearing potential(WCBP)† must have negative serum or urine pregnancy test 10 to 14 days prior to starting therapy. Patients with reproductive potential must use an adequate contraceptive method during treatment and for 3 months after completing treatment. In addition, sexually active WCBP must agree to use adequate contraceptive methods per the requirements outlined in protocol document.
* Patients treated with local radiotherapy with or without concomitant exposure to steroids, for pain control or management of cord/nerve root compression, are eligible. 4 weeks must have lapsed since last date of radiotherapy. Patients who require concurrent radiotherapy should have entry to the protocol deferred until radiotherapy is completed and 4 weeks have passed since last date of therapy.

Exclusion Criteria:

* Ongoing severe infection requiring intravenous antibiotic treatment
* Life expectancy < 3 months
* Prior malignancy, except; adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, or other cancer from which the participant has been disease-free for at least 5 years. Concurrent prostate cancer for which patient is receiving therapy will not be considered an exclusion if prostatic specific antigen (PSA) has been stable for 3 years.
* Solitary bone or solitary extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia
* Patients receiving therapeutic dosages of steroids for multiple myeloma
* Myocardial infarct within 6 months before enrollment, New York Heart Association (NYHA) Class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities
* Uncontrolled medical problems such as diabetes mellitus, coronary artery disease, hypertension, unstable angina, arrhythmias, pulmonary, hepatic and renal diseases unless renal insufficiency is felt to be secondary to multiple myeloma
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the informed consent form
* Pregnant or breast-feeding females. Lactating females must agree not to breast-feed.
* Any condition, including the presence of laboratory abnormalities, which places the participant at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Prior chemotherapy for multiple myeloma, except for radiation to symptomatic bony disease, plasmapheresis for hyperviscosity, kyphoplasty and/or vertebroplasty
* History of hypersensitivity reactions attributed to a conventional formulation of doxorubicin hydrochloride (HC1) or the components of DOXIL®
* Prior anthracycline dose exceeding 360 mg/m² for doxorubicin (including DOXIL) or 720 mg/m² for epirubicin
* Grade 2 or higher peripheral neuropathy on clinical examination within 14 days before enrollment
* Polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome or plasma cell leukemia
* Hypersensitivity to bortezomib, boron or mannitol
* Has received other investigational drugs within 14 days before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-09; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Alsina, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Moffitt Cancer Center from September 2008 to August 2011.
Groups:
- A. Phase I - Dose Escalation: Dose of Cyclophosphamide depended on how many patients we had treated. Three participants were treated at each level:
  * Dose Level 1: Cyclophosphamide 250 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Dose Level 2: Cyclophosphamide 500 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Dose Level 3: Cyclophosphamide 750 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Dose Level 4: Cyclophosphamide 750 mg /m^2 IV Day 1; VELCADE, 1.3 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
Period: Overall Study
Arm/Group | A. Phase I - Dose Escalation | B. Phase II - Maximum Planned Dose (MPD)
Started | 12 | 46
Completed | 12 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall Survival by disease risk stratification: 54 participants with cytogenetics and fluorescence in situ hybridisation (FISH) results available for risk stratification. All other measures: 58 Participants.
Groups:
- A. Phase I - Dose Escalation: Dose of Cyclophosphamide depended on how many patients we had treated:
  * Dose Level 1: Cyclophosphamide 250 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Dose Level 2: Cyclophosphamide 500 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Dose Level 3: Cyclophosphamide 750 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Dose Level 4: Cyclophosphamide 750 mg /m^2 IV Day 1; VELCADE, 1.3 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
- B. Phase II - Maximum Planned Dose (MPD): Participants received Cyclophosphamide and VELCADE at the MPD at the same schedule of the Phase I study. Pegylated doxorubicin and Dexamethasone were given at the same doses and schedule as the Phase I part of study.
- Total: Total of all reporting groups
Arm/Group | A. Phase I - Dose Escalation | B. Phase II - Maximum Planned Dose (MPD) | Total
Number analyzed (Participants) | 12 | 46 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 34 | 42
  >=65 years | 4 | 12 | 16
Age, Continuous [Mean (Full Range); unit: years] | 58.75 [46 to 77] | 57 [25 to 75] | 57 [25 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 20 | 24
  Male | 8 | 26 | 34
Region of Enrollment [Number; unit: participants]
  United States | 12 | 46 | 58

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Maximum Planned Dose (MPD) Level
Description: Maximum Phase II planned dose of cyclophosphamide when given in combination with bortezomib, pegylated liposomal doxorubicin and Dexamethasone (CVDD) in participants with newly diagnosed active multiple myeloma. Dose levels 1, 2, 3, 4 as outlined in Treatment Arm A.
  If no dose limiting toxicity (DLT) was reported in the first 3 participants at a dose level, that dose level was to be considered safe and 3 participants would be enrolled at the next dose level. If 1/3 participants in a cohort at a dose level had dose limiting toxicity (DLT), the dose level would be expanded to obtain 6 evaluable participants. MPD reflects the highest dose of drug that did not cause a DLT in 33% of participants.
Time Frame: 9 months
Population: All participants in Arm A. Three participants at each dose level.
Measure: Number; unit: Dosing Level
Groups:
- A. Phase I Dose Escalation: Dose of Cyclophosphamide depended on how many patients we had treated. Three participants were treated at each level:
  * Dose Level 1: Cyclophosphamide 250 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Dose Level 2: Cyclophosphamide 500 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Dose Level 3: Cyclophosphamide 750 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Dose Level 4: Cyclophosphamide 750 mg /m^2 IV Day 1; VELCADE, 1.3 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
Arm/Group | A. Phase I Dose Escalation
Number analyzed (Participants) | 12
Dosing Level | 4

2. Primary Outcome: Phase II: Overall Response Rate (ORR)
Description: Best response to CVDD chemotherapy. Overall Response: Partial Response (PR) + Very Good Partial Response (VGPR) + Complete Response (CR). PR: ≥ 50% reduction of serum M-protein and reduction in 24 hour urinary M-protein by ≥ 90% or to < 200 mg per 24 hours; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein with urine M-protein level < 100 mg per 24 hours; CR: Negative immunofixation on the serum and urine, disappearance of any soft tissue plasmacytomas, and ≤ 5% plasma cells in bone marrow.
Time Frame: Up to 6 months
Population: All Participants with Partial Response, Very Good Partial Response, or Complete Response.
Measure: Number; unit: participants
Groups:
- All Participants: Arm A:
  * Dose Level 1: Cyclophosphamide 250 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Dose Level 2: Cyclophosphamide 500 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Dose Level 3: Cyclophosphamide 750 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Dose Level 4: Cyclophosphamide 750 mg /m^2 IV Day 1; VELCADE, 1.3 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  Arm B:
  Participants received Cyclophosphamide and VELCADE at Level 4 (the MPD) at the same schedule of the Phase I study. Pegylated doxorubicin and Dexamethasone were given at the same doses and schedule as the Phase I part of study.
Arm/Group | All Participants
Number analyzed (Participants) | 54
participants
  Participants with Partial Response | 16
  Participants with Very Good Partial Response | 23
  Participants with Complete Response | 15

3. Secondary Outcome: Phase II: Progression-Free Survival (PFS)
Description: Progression-free survival after CVDD in participants with newly diagnosed active multiple myeloma. PFS: time from the initiation of therapy to progression, relapse or death from any causes.
  Progressive Disease (PD): Progressive Disease requires any one or more of the following:
  Increase of ≥ 25% from baseline in:
  * serum M-component and /or (the absolute increase must be ≥ 0.5 g/dL)
  * urine M-component and/or (the absolute increase must be ≥ 200 mg/24 h)
Time Frame: Up to 50.9 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Participants
Number analyzed (Participants) | 58
months | 31.3 [24.5 to NA] — Has not been reached

4. Secondary Outcome: Phase II: Two Year Overall Survival (OS)
Description: Overall survival by disease risk stratification after CVDD. OS: time from initiation of therapy until death from any cause.
Time Frame: 2 years
Population: Participants with cytogenetics and fluorescence in situ hybridisation (FISH) results available for risk stratification.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- High-Risk Myeloma: Participants eligible for risk stratification with High-Risk Myeloma.
  Arm A:
  * Level 1: Cyclophosphamide 250 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Level 2: Cyclophosphamide 500 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Level 3: Cyclophosphamide 750 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Level 4: Cyclophosphamide 750 mg /m^2 IV Day 1; VELCADE, 1.3 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  Arm B:
  Cyclophosphamide and VELCADE at Level 4 (the MPD) at the same schedule of the Phase I study. Pegylated doxorubicin and Dexamethasone were given at the same doses and schedule as Arm A.
- Standard-Risk Myeloma: Participants eligible for risk stratification with Standard-Risk Myeloma.
  Arm A:
  * Level 1: Cyclophosphamide 250 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Level 2: Cyclophosphamide 500 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Level 3: Cyclophosphamide 750 mg /m^2 IV Day 1; VELCADE, 1.0 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  * Level 4: Cyclophosphamide 750 mg /m^2 IV Day 1; VELCADE, 1.3 mg/m^2 IV days 1,4,8, and 11; DOXIL 30 mg/m^2 Day 4; Dexamethasone 20 mg orally daily on days 1-2,4-5,8-9,11-12
  Arm B:
  Cyclophosphamide and VELCADE at Level 4 (the MPD) at the same schedule of the Phase I study. Pegylated doxorubicin and Dexamethasone were given at the same doses and schedule Arm A.
Arm/Group | High-Risk Myeloma | Standard-Risk Myeloma
Number analyzed (Participants) | 12 | 42
percentage of participants | 88.9 [43.3 to 98.4] | 91.1 [78.0 to 96.6]

ADVERSE EVENTS:
Time Frame: Up to 6 months per participant
Groups:
- Dose Level 1: Participants at Dose Level 1
- Dose Level 2: Participants at Dose Level 2
- Dose Level 3: Participants at Dose Level 3
- Maximum Tolerated Dose: Participants at Dose Level 4
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Maximum Tolerated Dose
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 0/3 | 18/49
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=3) | Maximum Tolerated Dose (N=49)
Low Hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Low Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Low Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (in the absence of neutropenia) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection - Other (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Urinary tract NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Vulva (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infection with unknown ANC - Lymphatic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema: limb (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mental status (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (fainting) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pain - Other - rib cage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal/Genitourinary - Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=3) | Maximum Tolerated Dose (N=49)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 | 0 | 0 | 34
Insomnia (General disorders) | 0 | 0 | 1 | 20
Sweating (diaphoresis) (General disorders) | 0 | 0 | 0 | 17
Fever (in the absence of neutropenia) (General disorders) | 0 | 0 | 1 | 11
Rigors/chills (General disorders) | 0 | 0 | 0 | 11
Constitutional Symptoms - Other (General disorders) | 0 | 0 | 0 | 8
Weight Loss (General disorders) | 0 | 0 | 0 | 4
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 36
Low Platelets (Blood and lymphatic system disorders) | 0 | 1 | 0 | 29
Low Hemoglobin (Blood and lymphatic system disorders) | 0 | 0 | 0 | 27
Low Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 25
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 28
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 25
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 16
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 15
Gastrointestinal - Other (Gastrointestinal disorders) | 0 | 0 | 0 | 15
Anorexia (Gastrointestinal disorders) | 0 | 0 | 1 | 13
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 0 | 0 | 0 | 14
Dehydration (Gastrointestinal disorders) | 0 | 0 | 0 | 10
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 9
Distension/bloating, abdominal (Gastrointestinal disorders) | 0 | 0 | 0 | 5
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Neuropathy: sensory (Nervous system disorders) | 0 | 0 | 0 | 38
Dizziness (General disorders) | 0 | 0 | 0 | 20
Syncope (fainting) (General disorders) | 0 | 0 | 0 | 9
Mood alteration - Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 8
Neuropathy: motor (Nervous system disorders) | 0 | 0 | 0 | 6
Mood alteration - Depression (Psychiatric disorders) | 0 | 0 | 0 | 4
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 3
Mood alteration - Agitation (Psychiatric disorders) | 0 | 0 | 0 | 3
Tremor (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 21
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 12
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 9
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 6
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3
Rash: erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4
Flushing (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Rash: dermatitis associated with radiation - Chemoradiation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Pain - Other (General disorders) | 0 | 0 | 0 | 14
Pain - Head/headache (General disorders) | 0 | 0 | 0 | 13
Pain - Chest wall (General disorders) | 0 | 0 | 0 | 8
Pain - Back (General disorders) | 0 | 0 | 0 | 7
Pain - Extremity-limb (General disorders) | 0 | 0 | 1 | 6
Pain - Abdomen NOS (General disorders) | 0 | 0 | 0 | 5
Pain - Bone (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Pain - Neck (General disorders) | 0 | 0 | 0 | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 14
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 17
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 6
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3
Edema: limb (Blood and lymphatic system disorders) | 0 | 0 | 0 | 25
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 9
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 | 1 | 0 | 5
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 5
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 0 | 0 | 5
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 10
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 7
Hypotension (Cardiac disorders) | 0 | 0 | 0 | 13
Infection - Other (Infections and infestations) | 0 | 0 | 0 | 4
Febrile neutropenia (Infections and infestations) | 0 | 0 | 0 | 3
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1 | 0 | 0 | 2
Vision-blurred vision (Eye disorders) | 0 | 1 | 0 | 8
Ocular/Visual - Other (Eye disorders) | 0 | 0 | 0 | 4
Allergic rhinitis (Immune system disorders) | 0 | 0 | 0 | 8
Auditory/Ear - Other (Ear and labyrinth disorders) | 0 | 0 | 0 | 7
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 3
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 3
Hemorrhage/Bleeding - Other (General disorders) | 0 | 0 | 0 | 4
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 | 0 | 0 | 5
Renal/Genitourinary - Other (Renal and urinary disorders) | 0 | 0 | 0 | 3
Flu-like syndrome (General disorders) | 0 | 0 | 0 | 3

LIMITATIONS AND CAVEATS:
Trial closed early after 58 patients were enrolled due to slow accrual and shortage of pegylated liposomal doxorubicin. Only 54 participants had cytogenetics and fluorescence in situ hybridisation (FISH) results available for risk stratification.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes